CLINICAL TRIAL: NCT07108504
Title: An Open-label, Phase II Clinical Study to Evaluate the Efficacy and Safety of LM-302 Combined With Gemcitabine as Second-line Treatment for CLDN 18.2 Positive Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Efficacy and Safety of LM-302 Combined With Gemcitabine CLDN 18.2 Positive Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Liang Liu, Professor of Pancreatic Surgery, Zhongshan Hospital, Fudan University, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-16
Record Dates: First submitted 2025-07-30; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Chemotherapy Effect
Keywords: pancreatic adenocarcinoma; CLDN18.2; LM302; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LM-302 combined with Gemcitabine (Experimental)
  Interventions: Drug: Gemcitabine; Drug: LM-302

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine, 1000 mg/m², d1, 8, 15, q4 week
Drug: LM-302 — LM-302, 1.8 mg/kg, d1, q2 week

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of LM-302 combined with gemcitabine as a second-line treatment for CLDN 18.2-positive unresectable locally advanced or metastatic pancreatic cancer.

The main questions it aim to answer:

1. Does LM-302 plus gemcitabine improve the objective response rate (ORR, per RECIST 1.1) compared to historical controls?
2. What is the safety and tolerability profile of this combination therapy?

Participants will receive:

1. Gemcitabine (1000 mg/m² IV on Days 1, 8, and 15) in 4-week cycles, and LM-302 (1.8 mg/kg IV on Day 1) in 2-week cycles,
2. Undergo regular tumor imaging (CT/MRI) and safety assessments;
3. Provide blood samples for biomarker and pharmacokinetic analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written informed consent, understanding and complying with study requirements. Willing to participate after full disclosure of the study's purpose, procedures, potential risks, and benefits, and must sign the informed consent form before any study-related procedures.
2. Age ≥18 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, with no deterioration within 2 weeks before the first dose.
4. Expected survival ≥3 months.
5. Histologically or cytologically confirmed unresectable, locally advanced, or metastatic pancreatic ductal adenocarcinoma (PDAC) not amenable to curative treatment.
6. Must have experienced disease progression or intolerance to first-line standard therapy containing 5-FU (fluorouracil) (radiologically confirmed).
7. At least one measurable lesion per RECIST v1.1.
8. Must provide 5-7 unstained slides from archived (within 3 years) or fresh tumor tissue for CLDN18.2 and other biomarker testing. CLDN18.2 positivity defined as: Moderate-to-high staining intensity (2+~3+) in ≥50% of tumor cells, as assessed by central laboratory IHC (immunohistochemistry).
9. Adequate Organ Function (within 7 days before first dose) Bone marrow function: Platelets (PLT) ≥90 × 10⁹/L; Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; Hemoglobin ≥9 g/dL (no erythropoietin [EPO], G-CSF, or GM-CSF support within 14 days, and no transfusions within 7 days prior to treatment) Coagulation: INR ≤1.5; APTT ≤1.5 × ULN Liver function: Total bilirubin ≤1.5 × ULN (≤3 × ULN for Gilbert's syndrome); AST/ALT ≤2.5 × ULN (≤5 × ULN if liver metastases present); Serum albumin (ALB) ≥28 g/L Renal function: Serum creatinine ≤1.5 × ULN; Creatinine clearance (CrCl) ≥50 mL/min (calculated by Cockcroft-Gault formula) Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%; QTcF interval ≤470 ms
10. Females of childbearing potential and males with fertile partners must agree to use highly effective contraception from 7 days before the first dose until 6 months after the last dose.
11. Able to communicate effectively with investigators and comply with all study requirements.

Exclusion Criteria:

1. Previous treatment with gemcitabine or nab-paclitaxel.
2. Received any investigational drug or therapy within 28 days before the first dose of the study drug.
3. Recent Anticancer Therapy (within 21 days before the first dose, except for): Palliative radiotherapy (e.g., for bone metastasis pain control) within 14 days. Oral drugs (e.g., fluoropyrimidines, small-molecule targeted agents) within 14 days or 5 half-lives (whichever is longer). Traditional Chinese medicine with anticancer indications within 14 days. Nitrosoureas or mitomycin C within 42 days. Therapeutic radiopharmaceuticals within 56 days.
4. Residual Toxicities from Prior Therapy Adverse reactions from prior anticancer therapy have not recovered to CTCAE v5.0 Grade ≤1 (except for non-safety risks, such as alopecia, chronic radiotherapy toxicities ≤Grade 2, or lymphopenia).
5. Poorly Controlled Tumor-Related Pain Patients requiring analgesics must be on a stable dose before study entry.
6. Active or Untreated CNS Metastases Excludes those with previously treated, stable brain metastases (confirmed by imaging ≥4 weeks before the first dose, no new neurological symptoms, and no progression).
7. Proteinuria Urine protein ≥3+, or 2+ with 24-hour urine protein >1 g.
8. Recent Life-Threatening Hemorrhage Any major bleeding event within 3 months before the first dose.
9. High-Risk Esophageal/Gastric Varices Requires endoscopic evaluation within 3 months before the first dose if there is a history of variceal bleeding.
10. Severe Liver Dysfunction Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Class B/C cirrhosis.
11. Uncontrolled Third-Space Fluid Accumulation Clinically significant ascites/pleural effusion requiring repeated drainage, recent intervention (within 14 days), or causing complications (e.g., bowel obstruction).
12. Tumor Invasion of Critical Structures Encasement of major vessels (aorta, SVC, etc.) or risk of fistula formation (e.g., tracheoesophageal, pleuroesophageal).
13. History of GI Perforation/Fistula Within 6 months before the first dose.
14. Bowel Obstruction/Perforation Risk Complete/incomplete intestinal obstruction or high perforation risk within 3 months before the first dose.
15. Hypersensitivity to Antibody-Based Therapies History of ≥Grade 3 infusion reactions to monoclonal/bispecific antibodies, ≥Grade 3 immune-related AEs from prior immunotherapy, or discontinuation due to severe immune toxicity.
16. Recent Systemic Corticosteroid Use ≥10 mg/day prednisone (or equivalent) for >7 days within 2 weeks before the first dose (topical/ocular/inhaled steroids allowed).
17. Active Autoimmune Disease Includes but not limited to: Autoimmune hepatitis, SLE, rheumatoid arthritis, myasthenia gravis, multiple sclerosis. Exceptions: Stable hypothyroidism on hormone replacement, vitiligo, or psoriasis not requiring systemic therapy.
18. Inflammatory Bowel Disease (IBD) Active or history of Crohn's disease, ulcerative colitis, or chronic diarrhea.
19. Interstitial Lung Disease (ILD) Current or prior ILD requiring systemic corticosteroids.
20. Peripheral Neuropathy ≥Grade 2 sensory/motor neuropathy at screening.
21. Allergy to MMAE-Based ADCs Known ≥Grade 3 hypersensitivity to antibody-drug conjugates containing monomethyl auristatin E (MMAE).
22. Prior CLDN18.2-Targeted Therapy Any previous treatment targeting claudin 18.2 (CLDN18.2).
23. Strong CYP3A4 Modifiers Use of strong inhibitors/inducers within 14 days before the first dose.
24. Live Vaccination Received live/live-attenuated vaccines within 28 days (e.g., MMR, varicella, BCG, yellow fever). Allowed: Inactivated/mRNA COVID-19 vaccines, seasonal flu shots (non-nasal).
25. Therapeutic Anticoagulation Current use of heparin/warfarin (except prophylactic low-dose therapy).
26. Major Surgery/Trauma Undergone major surgery or invasive procedures within 28 days, or with unhealed wounds/fractures.
27. Severe Cardiovascular Disease Includes: Uncontrolled arrhythmias (e.g., ventricular tachycardia, AV block ≥Grade 2). Thromboembolism requiring anticoagulation. NYHA Class III/IV heart failure. Acute coronary syndrome, stroke, or ≥Grade 3 CV events within 6 months. Uncontrolled hypertension.
28. Active Infection Severe infections (e.g., sepsis, pneumonia) within 4 weeks, or ongoing systemic antibiotics within 2 weeks (except HBV/HCV antiviral therapy).
29. Immunodeficiency History of primary/secondary immunodeficiency, organ transplant, or stem cell transplant (unless no immunosuppression needed).
30. Chronic Viral Infections HIV-positive; Active HBV/HCV (exceptions): HBsAg+ if HBV DNA <500 IU/mL or undetectable; HCV Ab+ if HCV RNA negative.
31. Active Tuberculosis (TB) Must be ruled out clinically if suspected.
32. Other Malignancies Concurrent or history of other cancers within 5 years, except: Cured non-melanoma skin cancer, bladder CIS, low-risk prostate cancer (stage ≤T2a, Gleason ≤6, PSA ≤10 ng/mL), or cervical/breast CIS.
33. Pregnancy/Lactation Positive pregnancy test within 7 days or breastfeeding.
34. Psychiatric Disorders Conditions affecting compliance or safety judgment.
35. Non-Cancer-Related Systemic Illness Severe comorbidities (e.g., leukemoid reaction (WBC >20×10⁹/L), cachexia (>15% weight loss in 3 months).
36. Investigator's Discretion Any other condition deemed unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | From baseline until disease progression or study completion (up to 24 months).
  The proportion of participants with CLDN18.2-positive unresectable locally advanced or metastatic pancreatic adenocarcinoma achieving a best overall response of complete response (CR) or partial response (PR) as assessed by the investigator according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 | From first response until progression/death (up to 24 months).
  The time from first documented objective response (CR or PR) until disease progression or death, whichever occurs first, as assessed by RECIST 1.1.
Disease Control Rate (DCR) per RECIST 1.1 | From baseline until confirmed SD/response (up to 24 months).
  The proportion of participants achieving CR, PR, or stable disease (SD) lasting ≥16 weeks, as assessed by RECIST 1.1.
Progression-Free Survival (PFS) per RECIST 1.1 | From first dose of study treatment until disease progression (per RECIST 1.1) or death from any cause, assessed up to 24 months.
  Progression-Free Survival (PFS) is defined as the time from the first dose of study treatment (LM-302 + Gemcitabine) to the first occurrence of disease progression (per RECIST 1.1) or death from any cause, whichever occurs first.
Overall Survival (OS) | From first dose of study treatment until death from any cause or the end of follow-up, whichever occurs first, assessed up to 36 months.
  Overall Survival (OS) is defined as the time from the first dose of study treatment (LM-302 + Gemcitabine) to death from any cause.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose until 30 days after last dose (up to 24 months).
  Frequency and severity of adverse events (AEs), serious AEs (SAEs), and laboratory abnormalities graded by CTCAE v5.0.

IPD SHARING:
Plan to Share IPD: No